CLINICAL TRIAL: NCT04030468
Title: Effectiveness of Informative and/or Educational Interventions Aimed at Improving the Appropriate Use of Drugs Designed for General Practitioners and Their Patients
Brief Title: Educational and Informative Interventions to Tackle Inappropriate Use of Drugs in Italy
Acronym: EDUREDRUG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Milan (Other)
Collaborators: Federico II University (Other); University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Elena Tragni, Researcher at Epidemiology and Preventive Pharmacology Centre, University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FARM12KSBT; 2017-002622-21 (EudraCT Number)
Record Dates: First submitted 2019-07-19; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Inappropriate Drug Prescription and Use

STUDY DESIGN:
Intervention Model Description: According to the Local Health Unit (LHU), general practitioners (GPs) with their patients will be assigned to one of the following intervention arms:
  1. intervention on GPs (LHUs of Napoli 1 Nord and Bergamo)
  2. intervention on patients (LHUs of Avellino and Val Padana-Mantova District)
  3. intervention on GPs and patients (LHUs of Napoli 2 Centro and Brianza-Lecco District)
  4. no intervention (LHUs of Caserta and Brianza-Monza Brianza District)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- General practitioners (Experimental): Educational intervention
  Interventions: Other: Educational intervention addressed to general practitioners
- Patients (Experimental): Informative intervention
  Interventions: Other: Informative intervention addressed to patients
- General practitioners and patients (Experimental): Combined strategy
  Interventions: Other: Educational intervention addressed to general practitioners; Other: Informative intervention addressed to patients
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Educational intervention addressed to general practitioners — * feedback reports regarding the status of their patients according to the appropriateness indicators determined at baseline and the pooled prevalences for their patients, Local Health Units, and region
  * Continuous Medical Education (CME) course
  Arms: General practitioners; General practitioners and patients
Other: Informative intervention addressed to patients — • leaflets and posters distributed in primary care ambulatories and community pharmacies, focusing on correct drug use
  Arms: General practitioners and patients; Patients

SUMMARY:
Pharmacological intervention is an essential step in health promotion. However, lots of drugs are often used in inappropriate ways, especially in elderly patients. This study is aiming at evaluating the effectiveness of educational and/or informative interventions addressed to general practitioners and their adult patients in Italy, in order to improve appropriateness of prescribing in primary care.

DETAILED DESCRIPTION:
EDU.RE.DRUG project is a prospective, multicentre, open-label, parallel-arm, controlled, pragmatic trial directed to general practitioners (GPs) and their patients from two Italian regions (Campania and Lombardy), with the objective of investigating the practice of prescribing among GPs to highlight the most frequent events of inappropriateness and to implement ad hoc interventions for GPs and patients.

Appropriateness of prescribing in general practice will be assessed by evaluating selected prescribing, consumption and adherence indicators, using Regional administrative pharmaceutical prescription databases.

Primary care physicians and their patients will be assigned to four trial arms: informative intervention (leaflets and posters for patients), educational intervention (feedback reports and online CME courses for GPs), combined interventions, or no intervention. Intervention effectiveness will be assessed measuring the variation in rates of inappropriate prescription indicators after 1-year of follow-up.

EDU.RE.DRUG project will provide with improvements in the prescribing performance of GPs and in patients' adherence to treatment, with relevant clinical implications in terms of rational and safe use of drugs and optimized patient care, and with economic benefits (optimization of available resources use and savings in direct and indirect health costs).

ELIGIBILITY:
Inclusion Criteria:

* general practitioners of the Italian National Health System (NHS) operating at December 31, 2016 belonging to the 8 Local Health Units involved in the project

Exclusion Criteria:

* primary care pediatricians

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4840 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Inappropriate drug prescription and use indicators | 30 months
  Changes in prevalences of selected potentially inappropriate prescribing (including drug-drug interactions, duplicate therapies, inappropriate drugs in older people and drugs with high anticholinergic and sedative burden), consumption and adherence indicators between baseline and after the intervention

SECONDARY OUTCOMES:
Predictive factors of inappropriate prescribing | 30-36 months
  Identification of predictors of poor prescription appropriateness
Health Technology Assessment of intervention implemented | 30-36 months
  HTA analysis
GP's satisfaction | 30-36 months
  Level of general practitioners (GPs) satisfaction by using ad hoc web-based questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alberico L Catapano, Principal Investigator — University of Milan
Locations (1):
- SEFAP, University of Milan, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leendertse AJ, Egberts AC, Stoker LJ, van den Bemt PM; HARM Study Group. Frequency of and risk factors for preventable medication-related hospital admissions in the Netherlands. Arch Intern Med. 2008 Sep 22;168(17):1890-6. doi: 10.1001/archinternmed.2008.3. PMID 18809816
- [Background] Buetow SA, Sibbald B, Cantrill JA, Halliwell S. Appropriateness in health care: application to prescribing. Soc Sci Med. 1997 Jul;45(2):261-71. doi: 10.1016/s0277-9536(96)00342-5. PMID 9225413
- [Background] Spinewine A, Schmader KE, Barber N, Hughes C, Lapane KL, Swine C, Hanlon JT. Appropriate prescribing in elderly people: how well can it be measured and optimised? Lancet. 2007 Jul 14;370(9582):173-184. doi: 10.1016/S0140-6736(07)61091-5. PMID 17630041
- [Background] Goulding MR. Inappropriate medication prescribing for elderly ambulatory care patients. Arch Intern Med. 2004 Feb 9;164(3):305-12. doi: 10.1001/archinte.164.3.305. PMID 14769626
- [Background] Fialova D, Topinkova E, Gambassi G, Finne-Soveri H, Jonsson PV, Carpenter I, Schroll M, Onder G, Sorbye LW, Wagner C, Reissigova J, Bernabei R; AdHOC Project Research Group. Potentially inappropriate medication use among elderly home care patients in Europe. JAMA. 2005 Mar 16;293(11):1348-58. doi: 10.1001/jama.293.11.1348. PMID 15769968
- [Background] Maio V, Yuen EJ, Novielli K, Smith KD, Louis DZ. Potentially inappropriate medication prescribing for elderly outpatients in Emilia Romagna, Italy: a population-based cohort study. Drugs Aging. 2006;23(11):915-24. doi: 10.2165/00002512-200623110-00006. PMID 17109569
- [Background] Tragni E, Casula M, Pieri V, Favato G, Marcobelli A, Trotta MG, Catapano AL. Prevalence of the prescription of potentially interacting drugs. PLoS One. 2013 Oct 11;8(10):e78827. doi: 10.1371/journal.pone.0078827. eCollection 2013. PMID 24147143
- [Background] Beers MH, Ouslander JG, Rollingher I, Reuben DB, Brooks J, Beck JC. Explicit criteria for determining inappropriate medication use in nursing home residents. UCLA Division of Geriatric Medicine. Arch Intern Med. 1991 Sep;151(9):1825-32. PMID 1888249
- [Background] Casula M, Tragni E, Catapano AL. Adherence to lipid-lowering treatment: the patient perspective. Patient Prefer Adherence. 2012;6:805-14. doi: 10.2147/PPA.S29092. Epub 2012 Nov 8. PMID 23152673
- [Background] Thomas AN, Boxall EM, Laha SK, Day AJ, Grundy D. An educational and audit tool to reduce prescribing error in intensive care. Qual Saf Health Care. 2008 Oct;17(5):360-3. doi: 10.1136/qshc.2007.023242. PMID 18842975
- [Background] Ostini R, Hegney D, Jackson C, Williamson M, Mackson JM, Gurman K, Hall W, Tett SE. Systematic review of interventions to improve prescribing. Ann Pharmacother. 2009 Mar;43(3):502-13. doi: 10.1345/aph.1L488. Epub 2009 Mar 3. PMID 19261953
- [Background] Maio V, Del Canale S, Abouzaid S; GAP Investigators. Using explicit criteria to evaluate the quality of prescribing in elderly Italian outpatients: a cohort study. J Clin Pharm Ther. 2010 Apr;35(2):219-29. doi: 10.1111/j.1365-2710.2009.01094.x. PMID 20456742
- [Background] Husereau D, Drummond M, Petrou S, Carswell C, Moher D, Greenberg D, Augustovski F, Briggs AH, Mauskopf J, Loder E; ISPOR Health Economic Evaluation Publication Guidelines-CHEERS Good Reporting Practices Task Force. Consolidated Health Economic Evaluation Reporting Standards (CHEERS)--explanation and elaboration: a report of the ISPOR Health Economic Evaluation Publication Guidelines Good Reporting Practices Task Force. Value Health. 2013 Mar-Apr;16(2):231-50. doi: 10.1016/j.jval.2013.02.002. PMID 23538175